CLINICAL TRIAL: NCT04788472
Title: Clinical Trial for the Efficacy and Safety of Sequential CD19 and CD22 CAR-T Therapy for Adult Patients with Newly Diagnosed Ph Chromosome Positive B-cell Acute Lymphoblastic Leukemia
Brief Title: Sequential CD19 and CD22 CAR-T Therapy for Newly Diagnosed Ph+ B-ALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19-006
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: B-Cell Acute Lymphoblastic Leukemia, Adult
Keywords: CD19 CAR-T; CD22 CAR-T; Ph Chromosome Positive; B-ALL; Newly diagnosed
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T therapy (Experimental): Administration of CD19 and CD22 CAR T-cells
  Interventions: Drug: CAR-T cells targeting CD19 and CD22

INTERVENTIONS:
Drug: CAR-T cells targeting CD19 and CD22 — Each subject receives sequential CD19 and CD22 CAR-T cells by intravenous infusion

SUMMARY:
Clinical Trial for the Efficacy and Safety of Sequential CD19 and CD22 CAR-T Therapy for Adult Patients With Newly Diagnosed Ph Chromosome Positive B-cell Acute Lymphoblastic Leukemia

DETAILED DESCRIPTION:
This study was designed as a prospective, open-label, single-center study. It aims to evaluate the efficacy and safety of CD19 CAR-T cells in combination with dasatinib for the treatment of newly diagnosed Ph-positive B-cell acute lymphoblastic leukemia in adult.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Subjects with a diagnosis of B-cell acute lymphoblastic leukemia according to the 2016 edition of the WHO classification criteria for acute leukemia;
3. Subjects whose chromosomal and fusion gene analysis showed positivity for the Ph chromosome, BCR/ABL1 fusion gene;
4. Leukemia cells were CD19 and CD22 positive;
5. Patients with newly diagnosed B-ALL were not treated with standard chemotherapy regimens;
6. Serum total bilirubin ≤ 51 mol/L, serum ALT and AST both ≤ 3 times the upper limit of the normal range, blood creatinine ≤ 176.8 mol/L;
7. Echocardiography showed a left ventricular ejection fraction (LVEF) ≥50%;
8. Subjects had no active pulmonary infection and oxygen saturation ≥92% without oxygen;
9. The prognosis for survival is more than 3 months;
10. ECOG score 0-2;
11. Subjects volunteered to participate in this trial and signed an informed consent form.

Exclusion Criteria:

Subjects with any of the following exclusion criteria were not eligible for enrollment in this trial:

1. Those with a history of epilepsy or other central nervous system disorders;
2. Those with a history of prolonged QT period or severe cardiac disease;
3. Women who are pregnant or breastfeeding (the safety of this therapy for the unborn child is not known);
4. Those with uncontrolled active infection;
5. Active hepatitis B or hepatitis C virus infection;
6. Those who have previously used any gene therapy product;
7. Those with insufficient amplification (<5-fold) in response to CD3/CD28 co-stimulatory signals;
8. Creatinine > 2.5 mg/dl or ALT / AST > 3 times the upper limit of the normal range or bilirubin > 2.0 mg/dl;
9. Those who suffer from other uncontrolled medical conditions that, in the opinion of the investigator, make them unsuitable for enrollment;
10. HIV-infected persons;
11. Any condition that, in the opinion of the investigator, may increase the risk to the subject or interfere with the results of the test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Complete molecular response (CMR) rate | Up to 1 month after CAR-T cells infusion
  Complete molecular response (CMR) rate after CD19 CAR-T cell therapy

SECONDARY OUTCOMES:
Complete molecular response (CMR) rate | Up to 1 month after CAR-T cells infusion
  Complete molecular response (CMR) rate after CD22 CAR-T cell therapy
Leukemia-free survival (LFS) | Up to 2 years after CD19 CAR-T cells infusion
  From the complete remission to the occurrence of any event, including death, relapse (any one occurs first), and the last visit
Overall survival (OS) | Up to 2 years after CD19 CAR-T cells infusion
  From the first infusion of CD19 CAR-T cells to death or the last visit
cumulative incidence of relapse (CIR) | Up to 2 years after CD19 CAR-T cells infusion
  From the complete remission to relapse
Incidence of treatment-emergent adverse events (TEAEs) | Through study completion, an average of 2 years
  Incidence of treatment-emergent adverse events (Safety and Tolerability)
Characterization of relapse | Through study completion, an average of 2 years
  Including expression of CD19, CD22 and mutations in the ABL1 gene

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang M, Fu S, Feng J, Hong R, Wei G, Zhao H, Zhao M, Xu H, Cui J, Huang S, Wu X, Liu L, Sun J, Wu W, Zhu Y, He J, Zhao Y, Cai Z, Zheng W, Ye X, Shi J, Luo Y, Wang D, Chang AH, Hu Y, Huang H. Dasatinib and CAR T-Cell Therapy in Newly Diagnosed Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia: A Nonrandomized Clinical Trial. JAMA Oncol. 2025 Jun 1;11(6):625-629. doi: 10.1001/jamaoncol.2025.0674. PMID 40244598